CLINICAL TRIAL: NCT03711357
Title: Evaluation of the Effect of 980nm Diode Laser Intracanal Irradiation on Postoperative Pain and Root Canal Disinfection in Endodontic Retreatment Cases With Chronic Periapical Lesions
Brief Title: Effect of 980nm Diode Laser on Postoperative Pain and Root Canal Disinfection in Endodontic Retreatment Cases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Nabil El-Ezaby, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Eman Elezaby
Record Dates: First submitted 2018-10-13; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: A trial with two parallel groups
Who Masked: Participant
Masking Description: All the participants will be blinded, as they will not know which interventional group they belong to
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser (Active Comparator): 980 nm diode laser (maximum output of 3 watts and coupled with a fiber optic tip of 200 µm diameter) will be used for four irradiations, of 5 seconds each, after chemo-mechanical preparation procedures.
  Interventions: Radiation: 980 nm diode laser
- Placebo (Placebo Comparator): After chemo-mechanical preparation procedures, the diode laser fiber optic tip will be inserted inside the root canals but not activated.
  Interventions: Other: placebo

INTERVENTIONS:
Radiation: 980 nm diode laser — 980 nm high power diode laser device.
  Arms: laser
Other: placebo — the diode laser fiber optic tip will be inserted in root canals, but will not be activated.
  Arms: Placebo

SUMMARY:
A randomized clinical trial that evaluates the effect of using 980nm diode laser intracanal irradiation on postoperative pain and root canal disinfection in endodontic retreatment cases with chronic periapical lesions

DETAILED DESCRIPTION:
The endodontic retreatment procedures will be carried out for the participants, then 980nm Diode laser will be used to disinfect root canals. The researcher will then take microbiological samples of the root canals, to determine count and type of microorganisms in root canals. The subject will be asked to determine his level of pain at 7 days after endodontic retreatment procedures in a visual analogue scale (VAS), and to determine number of analgesic tablets needed to relieve his pain in the given charts. The subject will then return to the clinic 7 days later to bring back his charts. The researcher then will take another microbiological sample of the root canals, and complete the endodontic retreatment procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Endodontic retreatment cases of single rooted teeth with chronic periapical lesions; with periapical radiolucency of less than 1 cm diameter will be selected.
2. Teeth with straight root canals.
3. Subjects aged between 18-50 years of age.
4. No contributory medical history.
5. No previous administration of analgesics and / or antibiotics within the previous 2 weeks.

Exclusion Criteria:

1. Retreatment cases with complications such as separated instruments, perforations, ledges, resorption, transportation, calcifications, immature apices and over fillings.
2. Teeth with curved roots.
3. Swelling or sinus tract.
4. Mutilated teeth that interfere with proper isolation and seal between visits.
5. Subjects with generalized periodontitis, or if the tooth has probing depth of more than 3 mm.
6. Subjects with uncontrolled diabetes or debilitating diseases.
7. Pregnant or nursing females.
8. Systemic disorders that necessitate antibiotic prophylaxis or prevent the use of Ibuprofen.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
postoperative pain, measured using Visual analogue scale (VAS) | 7 days after root canal re-treatment procedures
  Visual analogue scale (VAS) will be used for to record severity of pain. It is a (0-10) scale. Criteria to determine the severity of postoperative pain will be as follows: (0: no pain), (1-3: mild pain), (4-6: moderate pain), (7-10: severe pain).

SECONDARY OUTCOMES:
Root canal disinfection | Four samples will be taken; first, second and third samples will be taken at first visit of endodontic retreatment procedures. while, the fourth sample will be taken in the second visit (7 days later).
  Number of microorganisms found in root canals will be determined using "Bacterial culture";"Initial sample", 'Pre-lasing sample, "Post-lasing". and "Recolonization sample", in the "Laser group" and "Placebo group".
number of analgesic tablets | At day 7 after endodontic retreatment procedures
  the participant will determine the number of analgesic tablets needed to relieve his pain after endodontic retreatment procedures.

IPD SHARING:
Plan to Share IPD: No
There is no plan to make the participants data available to other researchers